CLINICAL TRIAL: NCT02317432
Title: Building Community Capacity for Disability Prevention for Minority Elders
Brief Title: Building Community Capacity for Disability Prevention for Minority Elders (Positive Minds - Strong Bodies)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: New York University (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01AG046149-01A1 (NIH)
Record Dates: First submitted 2014-11-12; First posted 2014-12-16 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Depression; Anxiety; Physical Disability
Keywords: Depression; Anxiety; Disability; Ethnic Minority; Elders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT + InVEST exercise (Experimental): 10 sessions of individual CBT plus 36 sessions of InVEST group exercise, provided over a 12-week intervention period.
  Interventions: Behavioral: Comparison of a combined CBT + exercise intervention and enhanced usual care
- Enhanced Usual Care (Active Comparator): Usual care, as accessed through the community-based organization, plus written material from the NIH on depression, anxiety, and physical health for elders.
  Interventions: Behavioral: Comparison of a combined CBT + exercise intervention and enhanced usual care

INTERVENTIONS:
Behavioral: Comparison of a combined CBT + exercise intervention and enhanced usual care

SUMMARY:
The primary intervention offered through this study is a manualized and culturally adapted CBT intervention combined with an exercise intervention, administered by trained Community Health Workers and exercise trainers to ethnic minority elders with moderate to severe mood symptoms and at risk of disability. In addition to the intervention implementation, the study examines how to successfully build collaborative research for the provision of evidence-based mental health and disability prevention treatments for ethnic minority elders in community-based settings. Thus, the study will evaluate the three components necessary for a successful intervention: efficacy, since the intervention must work, acceptability among clients and partnering agencies, and feasibility and sustainability within the organization.

DETAILED DESCRIPTION:
The researchers have partnered with 5 community-based organizations and 2 clinics, each of whom will recruit 60 elder participants to be randomized into either the intervention (CBT+exercise) or control (enhanced usual care) groups. Each participant randomized into the intervention group will receive 10 sessions of individual CBT for depression and anxiety (Positive Minds), using a translated and culturally adapted manual, and administered by a trained community health worker. In addition, each participant will engage in three exercise groups per week for 12 weeks, using the Increased Velocity Specific to Task (Strong Bodies; InVEST) protocol. Both intervention and control groups will be assessed biweekly for symptoms of depression, anxiety, and suicidality, and both groups will participate in a thorough assessment at baseline, and 2, 6, and 12 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+
* Fluency in English, Spanish, Mandarin or Cantonese
* Score above threshold on PHQ-9, GAD-7, or Geriatric Depression Scale (GDS-Short Form)
* Score within threshold of SPPB

Exclusion Criteria:

* Participants will be excluded if there is evidence of:
* Current substance use disorders
* Current or last 3 months of specialty mental health treatment
* Evidence that patient the participant lacks capacity to consent assessed using the UCSD Brief Assessment of Capacity to Consent.
* Suicidal risk (score of 4 or 5 on the Paykel suicide questionnaire), whereby participant will be referred for immediate treatment to specialty care
* If the participant's physician advises against strenuous physical exercise.
* Exclusion from the disability component will also happen if the participant is home-bound, has an acute or an exacerbated chronic disease, or has neuro-musculoskeletal impairment that prevents them from participating in the exercises

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2015-07; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Alegria, PhD, Principal Investigator — Massachusetts General Hospital
Locations (8):
- United States (7):
  - King David Foundation, Aventura, Florida
  - Greater Boston Chinese Golden Age Center, Boston, Massachusetts
  - MGH Chelsea, Chelsea, Massachusetts
  - Kit Clark Senior Services, Dorchester, Massachusetts
  - MGH Revere, Revere, Massachusetts
  - Central Harlem Senior Citizens' Center, New York, New York
  - Hamilton Madison City Hall Senior Center, New York, New York
- University of Puerto Rico, San Juan, PR, Puerto Rico

REFERENCES:
- [Derived] Zhang L, Cruz-Gonzalez M, Lin Z, Ouyang X, Zhao F, Alegria M. Association of everyday discrimination with health outcomes among Asian and non-Asian US older adults before and during the COVID-19 pandemic. Front Public Health. 2022 Oct 19;10:953155. doi: 10.3389/fpubh.2022.953155. eCollection 2022. PMID 36339195
- [Derived] Porteny T, Alegria M, Del Cueto P, Fuentes L, Markle SL, NeMoyer A, Perez GK. Barriers and strategies for implementing community-based interventions with minority elders: positive minds-strong bodies. Implement Sci Commun. 2020 Apr 30;1:41. doi: 10.1186/s43058-020-00034-4. eCollection 2020. PMID 32885198

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care
Started | 153 | 154
Completed CBT (Completed 50% or more (5 or more) Positive Minds CBT sessions, which is considered the appropriate threshold for populations not recognizing the need for services and not actively seeking treatment.) | 118 | 0 (Participants in Enhanced Usual Care did not receive CBT sessions.)
Completed InVEST (Completed 50% or more (18 or more) Strong Minds InVEST sessions, which is considered the appropriate threshold for populations not recognizing the need for services and not actively seeking treatment.) | 63 | 0 (Participants in Enhanced Usual Care did not receive InVEST sessions.)
Completed CBT + InVEST Exercise (Completed either 50% or more Positive Minds CBT sessions or 50% or more Strong Minds InVEST sessions.) | 122 | 0 (Participants in Enhanced Usual Care did not receive either CBT or InVEST sessions.)
Completed Enhanced Usual Care | 0 (Participants in CBT + InVEST exercise did not receive Enhanced Usual Care.) | 148
Completed | 122 | 148
Not Completed | 31 | 6
Not completed — Death | 4 | 1
Not completed — Lost to Follow-up | 0 | 5
Not completed — Did not complete any CBT/InVEST sessions or the recommended number of sessions | 27 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care | Total
Number analyzed (Participants) | 153 | 154 | 307
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 144 | 142 | 286
Age, Continuous [Mean (Full Range); unit: years] | 74.86 [62 to 94] | 75.44 [62 to 95] | 75.15 [62 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 125 | 248
  Male | 30 | 29 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 72 | 136
  Not Hispanic or Latino | 64 | 55 | 119
  Unknown or Not Reported | 25 | 27 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 6 | 8
  Asian | 51 | 51 | 102
  Native Hawaiian or Other Pacific Islander | NA — The race was not an option when collecting data. | NA — The race was not an option when collecting data. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 15 | 14 | 29
  White | 50 | 47 | 97
  More than one race | 26 | 30 | 56
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 153 | 154 | 307
Hopkins Symptom Checklist-25 (HSCL-25) [Mean (Standard Deviation); unit: units on a scale] — The HSCL-25 is a 25-item screener of mood symptoms (ten anxiety symptoms and 15 depressive symptoms). Respondents are asked how much they were bothered by each symptom in the last four weeks, with responses rated on a 4-point scale (1 = not at all and 4 = extremely). Total scores are computed averaging all items (range: 1-4), and higher scores represent worse symptoms.
  units on a scale | 1.62 (.42) | 1.63 (.46) | 1.62 (.44)
Short Physical Performance Battery (SPPB) [Mean (Standard Deviation); unit: units on a scale] — The SPPB is an assessment tool developed by the National Institute of Aging to evaluate lower extremity functioning in older persons. It includes three tests (subscales) of functional relevance: standing balance, 4-meter gait speed, and five-repetition sit-to-stand motion. Each of the three components is scored on a 5-point subscale from 0 (unable to perform or low performance) to 4 (high performance). These three subscales are added to obtain a summary score than ranges between 0 and 12, with higher scores representing higher performance of physical functioning.
  units on a scale | 7.58 (2.30) | 7.38 (2.03) | 7.48 (2.17)
Function Component of the Late Life Functioning and Disability Instrument (LLFDI) [Mean (Standard Deviation); unit: units on a scale] — The function component of the LLFD is a 32-item self-reported measure assessing difficulty in performing discrete daily physical activities in older adults. Respondents are asked about difficulties performing an activity without help from someone else or the use of assisted devices, with responses rated on a 5-point scale (1 = cannot do and 5 = none). Total scores are calculated summing all items (range: 32-160), and scores approaching 32 indicate poor ability.
  units on a scale | 118.42 (25.96) | 116.75 (26.20) | 117.58 (26.05)
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) [Mean (Standard Deviation); unit: units on a scale] — The WHODAS 2.0 is a 12-item measure of level of functioning in six domains of life: Cognition, mobility, self-care, getting along, life activities, and participation. Respondents are asked about functioning difficulties experienced in the last 30 days, with responses rated on a 5-point scale (1 = none and 5 = extreme or cannot do). Final scores are calculated summing all items (range: 12-60), and higher scores represent more difficulties.
  units on a scale | 21.97 (7.09) | 22.40 (7.86) | 22.19 (7.48)
Generalized Anxiety Disorder 7-item Scale (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — The GAD-7 is a 7-item self-reported tool to identify probable cases of Generalized Anxiety Disorder. Respondents are asked how often, during the last two weeks, they were bothered by each symptom, with responses rated on a 4-point scale (0 = not at all and 3 = nearly every day). Total scores are calculated summing all items (range: 0-21), and higher scores represent worse symptoms.
  units on a scale | 6.18 (4.63) | 5.79 (4.56) | 5.99 (4.59)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending More Than 50% of Intervention Sessions and Number of Participants Reporting Satisfaction With the Intervention Sessions
Description: The number of participants attending more than 50% of intervention sessions was measured in three ways: (1) number attending 50% or more of the CBT sessions (CBT), (2) number attending 50% or more of the InVEST exercise sessions (InVEST), and (3) number attending 50% or more of the CBT and InVEST sessions (CBT and InVEST). Satisfaction with the intervention sessions was measured as the number of participants reporting to be "very satisfied".
Time Frame: 6-months post-baseline
Population: Analysis population includes only participants in the CBT + InVEST exercise group because the outcome (number of participants attending more than 50% of the intervention sessions and reporting satisfaction with the intervention sessions) cannot be measured for participants in the Enhanced Usual Care group since they did not receive the intervention sessions.
Measure: Count of Participants; unit: Participants
Groups:
- CBT + InVEST Exercise: 10 sessions of individual CBT plus 36 sessions of InVEST group exercise, provided over a 12-week intervention period.
  Comparison of a combined CBT + exercise intervention and enhanced usual care
- Enhanced Usual Care: Usual care, as accessed through the community-based organization, plus written material from the NIH on depression, anxiety, and physical health for elders.
  Comparison of a combined CBT + exercise intervention and enhanced usual care
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care
Number analyzed (Participants) | 153 | 0
Participants
  CBT | 118 |
  InVEST | 63 |
  CBT and InVEST | 58 |
  Satisfaction (very satisfied) | 121 |

2. Primary Outcome: Change in Mood Symptoms in the Hopkins Symptom Checklist-25 (HSCL-25) From Baseline, at 6-month Follow-up
Description: The HSCL-25 is a 25-item screener of mood symptoms (ten anxiety symptoms and 15 depressive symptoms). Respondents are asked how much they were bothered by each symptom in the last four weeks, with responses rated on a 4-point scale (1 = not at all and 4 = extremely). Total scores are computed averaging all items (range: 1-4), and higher scores represent worse symptoms.
Time Frame: 6-months post-baseline
Population: Intent to treat population (all participants assigned to CBT + InVEST exercise or Enhanced Usual Care). Multiple imputation by chained equations (MICE) imputation method.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care
Number analyzed (Participants) | 153 | 154
units on a scale | 1.44 (.030) | 1.56 (.038)
Statistical Analysis 1: Comparison: CBT + InVEST Exercise vs Enhanced Usual Care; Test type: Superiority; p < 0.01, Mixed Models Analysis — Threshold for statistical significance was p<0.05; Slope = -0.12

3. Primary Outcome: Change in Functional Limitations in the Short Physical Performance Battery (SPPB) From Baseline, at 6-month Follow-up
Description: The SPPB is an objective assessment tool developed by the National Institute of Aging to evaluate lower extremity functioning in older persons. It includes three tests (subscales) of functional relevance: standing balance, 4-meter gait speed, and five-repetition sit-to-stand motion. Each of the three components is scored on a 5-point subscale from 0 (unable to perform or low performance) to 4 (high performance). These three subscales are added to obtain a summary score than ranges between 0 and 12, with higher scores representing higher performance of physical functioning.
Time Frame: 6-months post-baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care
Number analyzed (Participants) | 153 | 154
units on a scale | 7.89 (0.22) | 7.29 (0.19)
Statistical Analysis 1: Comparison: CBT + InVEST Exercise vs Enhanced Usual Care; Test type: Superiority; p = 0.03, Mixed Models Analysis — Threshold for statistical significance was p<0.05; Slope = 0.60

4. Primary Outcome: Change in Self-reported Level of Functioning in the Function Component of the Late Life Functioning and Disability Instrument (LLFDI) From Baseline, at 6-month Follow-up.
Description: The Function Component of the LLFDI is a 32-item self-reported measure assessing difficulty in performing discrete daily physical activities in older adults. Respondents are asked about difficulties performing an activity without help from someone else or the use of assisted devices, with responses rated on a 5-point scale (1 = cannot do and 5 = none). Total scores are calculated summing all items (range: 32-160), and lower scores (approaching 32) are worse as they indicate more difficulties performing discrete daily activities, while higher scores are better as they indicate less difficulties.
Time Frame: 6-months post-baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care
Number analyzed (Participants) | 153 | 154
units on a scale | 120.87 (2.34) | 114.87 (2.16)
Statistical Analysis 1: Comparison: CBT + InVEST Exercise vs Enhanced Usual Care; Test type: Superiority; p = 0.02, Mixed Models Analysis — Threshold for statistical significance was p<0.05; Slope = 6.00

5. Primary Outcome: Change in Level of Functioning in the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) From Baseline, at 6-month Follow-up.
Description: The WHODAS 2.0 is a 12-item measure of level of functioning in six domains of life: Cognition, mobility, self-care, getting along, life activities, and participation. Respondents are asked about functioning difficulties experienced in the last 30 days, with responses rated on a 5-point scale (1 = none and 5 = extreme or cannot do). Final scores are calculated summing all items (range: 12-60), and higher scores represent more difficulties.
Time Frame: 6-months post-baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care
Number analyzed (Participants) | 153 | 154
units on a scale | 21.23 (0.66) | 22.47 (0.69)
Statistical Analysis 1: Comparison: CBT + InVEST Exercise vs Enhanced Usual Care; Test type: Superiority; p = 0.15, Mixed Models Analysis — Threshold for statistical significance was p<0.05; Slope = -1.24

6. Primary Outcome: Change in Anxiety Symptoms in the Generalized Anxiety Disorder 7-item Scale (GAD-7) From Baseline, at 6-month Follow-up
Description: The GAD-7 is a 7-item self-reported tool to identify probable cases of Generalized Anxiety Disorder. Respondents are asked how often, during the last two weeks, they were bothered by each symptom, with responses rated on a 4-point scale (0 = not at all and 3 = nearly every day). Total scores are calculated summing all items (range: 0-21), and higher scores represent worse symptoms.
Time Frame: 6-moths post-baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care
Number analyzed (Participants) | 153 | 154
units on a scale | 4.80 (0.38) | 5.29 (0.39)
Statistical Analysis 1: Comparison: CBT + InVEST Exercise vs Enhanced Usual Care; Test type: Superiority; p = 0.35, Mixed Models Analysis — Threshold for statistical significance was p<0.05; Slope = -0.49

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | CBT + InVEST Exercise | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 4/153 | 1/154
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/154
Other Adverse Events (participants affected / at risk) | 0/153 | 0/154

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT02317432/Prot_SAP_000.pdf